CLINICAL TRIAL: NCT00190060
Title: Study of The Effects of Testosterone on Muscle Function, Physical Performance, Body Composition and Quality of Life in Frail Elderly Men
Brief Title: Study of The Effects of Testosterone in Frail Elderly Men
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: University of Manchester (Other); Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMMCHUT PIN 9197; T0053/WTCRF
Record Dates: First submitted 2005-09-11; First posted 2005-09-19 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Frailty; Sarcopenia
Keywords: Frailty; Muscle strength; Physical performance; Bone mineral density; Quality of life
MeSH Terms: conditions — Frailty; Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Transdermal testosterone gel (Testogel 1% )
  Interventions: Drug: Transdermal testosterone gel (Testogel 1% )
- 2 (Placebo Comparator): Matched transdermal placebo gel
  Interventions: Drug: Matched transdermal placebo gel

INTERVENTIONS:
Drug: Transdermal testosterone gel (Testogel 1% ) — Transdermal testosterone gel (Testogel 1% ), 50 mg/d for 6 months
  Other Names: Testogel 1%
  Arms: 1
Drug: Matched transdermal placebo gel — Matched transdermal placebo gel, 50mg/d for 6 months
  Arms: 2

SUMMARY:
The study aims to determine the effects of testosterone on muscle function, mobility, activities of daily living and overall quality of life

DETAILED DESCRIPTION:
Ageing-associated loss of muscle mass and strength is a major cause of physical frailty, disability, morbidity and dependency in the elderly. This is associated with increased falls, fractures, loss of mobility, restricted activities of daily living and increased utilisation of healthcare resources. It is well known that serum testosterone levels fall with advancing age and this may be an important cause for muscle wasting and weakness (sarcopenia). Testosterone replacement increases muscle mass and improves muscle strength in young hypogonadal men. In relatively healthy elderly men, some short-term studies have also shown that testosterone can improve muscle strength. The potential beneficial effects of testosterone supplementation on muscle strength and functional capacity of frail elderly men has so far not been studies and forms the basis of this research. We hypothesise that testosterone supplementation is an effective, safe and economic anabolic intervention in frail elderly men with low circulating testosterone.

ELIGIBILITY:
Inclusion Criteria:

* Frail elderly men (as defined by Freid's criteria of frailty)
* Community - dwelling men aged 65 years and above
* Total testosterone ≤12.0 nmol/L or calculated free T≤0.25nmol/L

Exclusion Criteria:

* Carcinoma of prostate
* Carcinoma of breast
* PSA >4ng/mL
* Severe symptomatic benign prostatic hypertrophy (IPSS >21)
* Active liver disease
* Renal impairment (serum creatinine >180 mmol/L)
* Congestive heart failure
* Unstable ischaemic heart disease
* Polycythaemia
* Evidence of systemic disease which may affect muscle/joint function
* Moderate to severe peripheral vascular disease
* Moderate to severe chronic obstructive airways disease
* Alcohol consumption over 30 units per week
* Medications that interfere with sex steroid metabolism
* History of stroke causing persistent motor deficit
* Cognitive deficit
* Major psychiatric illness
* Hospital admission in the past 6 weeks
* Sleep apnoea

Min Age: 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 262 (Actual)
Dates: Start 2004-10; Primary Completion 2008-12-31 (Actual); Study Completion 2008-12-31 (Actual)

PRIMARY OUTCOMES:
Lower limb muscle strength at 6 months | 6 months

SECONDARY OUTCOMES:
Upper limb muscle strength at 6 months | 6 months
Quality of life at 6 months | 6 months
Total and regional lean body mass at 6 months | 6 months
Improvement in physical performance | 6 months
Bone Mineral Density | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Professor Frederick CW Wu, MD, FRCP, Principal Investigator — Central Manchester and Manchester Children's University Hospitals Trust & The University of Manchester; Dr Martin Connolly, MD, FRCP, Principal Investigator — Central Manchester and Manchester Children's University Hospitals Trust; Professor JA Oldham, PhD, Principal Investigator — The University of Manchester
Locations (1):
- Wellcome Trust Clinical Research Facility, Manchester Royal Infirmary, Manchester, United Kingdom

REFERENCES:
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Deslypere JP, Vermeulen A. Leydig cell function in normal men: effect of age, life-style, residence, diet, and activity. J Clin Endocrinol Metab. 1984 Nov;59(5):955-62. doi: 10.1210/jcem-59-5-955. PMID 6480814
- [Background] Clague JE, Wu FC, Horan MA. Difficulties in measuring the effect of testosterone replacement therapy on muscle function in older men. Int J Androl. 1999 Aug;22(4):261-5. doi: 10.1046/j.1365-2605.1999.00177.x. PMID 10442299
- [Background] Bhasin S, Woodhouse L, Casaburi R, Singh AB, Bhasin D, Berman N, Chen X, Yarasheski KE, Magliano L, Dzekov C, Dzekov J, Bross R, Phillips J, Sinha-Hikim I, Shen R, Storer TW. Testosterone dose-response relationships in healthy young men. Am J Physiol Endocrinol Metab. 2001 Dec;281(6):E1172-81. doi: 10.1152/ajpendo.2001.281.6.E1172. PMID 11701431
- [Derived] O'Connell MD, Roberts SA, Srinivas-Shankar U, Tajar A, Connolly MJ, Adams JE, Oldham JA, Wu FC. Do the effects of testosterone on muscle strength, physical function, body composition, and quality of life persist six months after treatment in intermediate-frail and frail elderly men? J Clin Endocrinol Metab. 2011 Feb;96(2):454-8. doi: 10.1210/jc.2010-1167. Epub 2010 Nov 17. PMID 21084399